CLINICAL TRIAL: NCT07041944
Title: "Efficacy and Usability of HEMImprove 1.0 Gamified Mobile Application for Upper Limb Rehabilitation in Adolescents With Unilateral Cerebral Palsy: A Randomized Controlled Trial"
Brief Title: HEMImprove 1.0 in Children and Adolescents With Unilateral Cerebral Palsy
Acronym: HEMImprove-APP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEMImprove-APP; FEDER (Other: FEDER)
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Unilateral Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Use HEMImprove 1.0 mobile app at home for 30 minutes/session, 5 days/week, for 4 weeks. Exercises tailored progressively with avatar guidance.
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know the group where the child/adolescent is (experimental or control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEMImprove APP (Experimental): Experimental Group:
  Use HEMImprove 1.0 mobile app at home for 30 minutes/session, 5 days/week, for 4 weeks. Exercises tailored progressively with avatar guidance.
  Control Group:
  Perform conventional home exercises guided by printed manual with instructions and images, matching frequency and duration of intervention group.
  Interventions: Other: HEMImprove APP
- Control group (Active Comparator): The control group will do exercises for the same time that is described in the experimental group, without using the APP
  Interventions: Other: exercises to upper limb

INTERVENTIONS:
Other: HEMImprove APP — Experimental Group:
  Use HEMImprove 1.0 mobile app at home for 30 minutes/session, 5 days/week, for 4 weeks. Exercises tailored progressively with avatar guidance.
  Control Group:
  Perform conventional home exercises guided by printed manual with instructions and images, matching frequency and duration of intervention group.
  Arms: HEMImprove APP
Other: exercises to upper limb — The patients will do the same exercises than the experimental group, without APP and using the same dosage
  Arms: Control group

SUMMARY:
This study aims to evaluate the effectiveness and usability of HEMImprove 1.0, a gamified mobile application designed to improve upper limb motor function in adolescents with unilateral cerebral palsy. Participants will be randomly assigned to an intervention group using the app or a control group performing conventional home exercises. The intervention will last four weeks, with assessments before and after the intervention to measure motor function, motivation, and quality of life improvements.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 18 years diagnosed with unilateral cerebral palsy.
* Ability to use the mobile app independently or with minimal assistance.
* Informed consent provided.

Exclusion Criteria:

* Severe cognitive impairment.
* Recent upper limb surgery (within 6 months).
* Recent botulinum toxin treatment (within 3 months).
* Other neurological or orthopedic disorders affecting upper limb function.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment | baseline, immediately after the intervention, 3 months after intervention
Melbourne Assessment v 2.0 MA2 | baseline, immediately after the intervention, 3 months after intervention
Nine hole Test | baseline, immediately after the intervention, 3 months after intervention

SECONDARY OUTCOMES:
User satisfaction and usability measured through structured Likert-scale questionnaires post-intervention. | From the recruitment to the follow-up
Qualitative data from semi-structured interviews analyzing user experience. | from the recruitment to the end of the treatment